CLINICAL TRIAL: NCT00698399
Title: Serum Markers of Ischemia Reperfusion Injury in Liver Transplant Patients, Phase II
Brief Title: Serum Markers of Ischemia Reperfusion Injury in Liver Transplant Patients
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 80237
Record Dates: First submitted 2008-06-12; First posted 2008-06-17 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Liver Transplant
Keywords: liver; transplant; TMAO; NGAL; cystatin-C; Ischemia Reperfusion Injury; Liver Transplant; LTx; allantion
MeSH Terms: conditions — Reperfusion Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum of patients who are undergoing liver transplantation surgery
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Live Donor
- 2: Cadaveric Donor

SUMMARY:
This is an observational study examining serum markers in patients who are undergoing either a cadaveric liver transplant or a living related liver transplant.

DETAILED DESCRIPTION:
The Departments of Anesthesiology are conducting an observational trial of markers in the serum of patients who are undergoing liver transplantation surgery. This study will utilize the biological markers, trimethylamine-N-oxide (TMAO), NGAL, and cystatin-C, sensitive markers of renal medullary injury in the blood and allantoin, a marker of oxidative stress as indicators of renal injury in a kidney during liver transplants. It is hypothesized that: (1) these markers are less pronounced in living donor liver transplant recipient patients than in cadaveric liver transplant recipients, and (2) these markers are less pronounced in cadaveric liver transplant recipients in which a "piggy-back" technique was used versus recipients in which a total venous occlusion technique was used. This study will be done in a multi-center format, along with researchers at UCSF

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Class I-V.
* Patient is undergoing elective Liver Transplant Surgery.
* Patient is an adult, 18 years old or older.

Exclusion Criteria:

* Patients < 18 Years of Age
* Patients who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from those on the list awaiting liver transplantation at Vanderbilt University Medical Center (VUMC). They will be recruited by the investigators prior to the time of their transplantation surgery
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-03; Primary Completion 2010-02-02 (Actual); Study Completion 2010-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M Waldman, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- See also: Vanderbilt University Medical Center Department of Anesthesiology — http://www.vandydreamteam.com